CLINICAL TRIAL: NCT05564442
Title: Comparative Evaluation of Different Pain Alleviating Methods During Intra-oral Local Anesthetic Injections in Children : A Randomized Controlled Trial
Brief Title: Compare the Efficacy of Various Pain Alleviating Methods in Reducing Pain in Children During Intraoral Local Anaesthetic Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Bahy ibrahim abdelfatah ellmelegy, Principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 581/2022
Record Dates: First submitted 2022-08-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I: Children received 20% benzocaine gel (Active Comparator): Comparative Evaluation of Different Pain Alleviating Methods During Intra-oral Local Anesthetic Injections
  Interventions: Drug: 20% benzocaine gel
- Group II: Children received TENS stimuli (Active Comparator): Comparative Evaluation of Different Pain Alleviating Methods During Intra-oral Local Anesthetic Injections
  Interventions: Device: Transcutaneous electric nerve stimuli
- Group III: Children received EMLA gel. (Active Comparator): Comparative Evaluation of Different Pain Alleviating Methods During Intra-oral Local Anesthetic Injections
  Interventions: Drug: Emla gel
- Group IV: Children received ice application at injection site (Active Comparator): Comparative Evaluation of Different Pain Alleviating Methods During Intra-oral Local Anesthetic Injections
  Interventions: Other: Ice application

INTERVENTIONS:
Drug: 20% benzocaine gel — compare the efficacy of various pain alleviating methods by application of Emla gel, TENS, and topical cooling of injection sites with 20% benzocaine gel in children 6-10 years requiring anesthesia during routine dental procedures.
  Arms: Group I: Children received 20% benzocaine gel
Device: Transcutaneous electric nerve stimuli — compare the efficacy of various pain alleviating methods by application of Emla gel, TENS, and topical cooling of injection sites with 20% benzocaine gel in children 6-10 years requiring anesthesia during routine dental procedures.
  Arms: Group II: Children received TENS stimuli
Drug: Emla gel — compare the efficacy of various pain alleviating methods by application of Emla gel, TENS, and topical cooling of injection sites with 20% benzocaine gel in children 6-10 years requiring anesthesia during routine dental procedures.
  Arms: Group III: Children received EMLA gel.
Other: Ice application — compare the efficacy of various pain alleviating methods by application of Emla gel, TENS, and topical cooling of injection sites with 20% benzocaine gel in children 6-10 years requiring anesthesia during routine dental procedures.
  Arms: Group IV: Children received ice application at injection site

SUMMARY:
The aim of study is to compare the efficacy of various pain alleviating methods by application of Emla gel, TENS, and topical cooling of injection sites compared with 20% benzocaine gel in reducing pain in children requiring anesthesia during routine dental procedures.

DETAILED DESCRIPTION:
The main concern of the pediatric dentist is to achieve the cooperation of the child in the dental clinic during various pediatric procedures. Administering anesthesia to pediatric patients is the most challenging part of the process. The real fear of the child during a pediatric procedure is painful local anesthetic (LA) injections. The mere sight of needle and syringes cause psychological trauma to the child and thus interferes with the behavior management of a child. Reducing the fear of pain during LA injections gains the confidence of the child toward the dentist, thus achieving the cooperation of the child during treatment .

To reduce the pain during administration of the LA injection, several pharmacological and non-pharmacological methods such as use of topical anesthetics, slowing down the rate of infiltration, distracting the children, vibrating the tissue of the injection site during injection, heat and ice application before the injection have been tested. Application of flavored topical anesthetic gel is most commonly practiced in pediatric dentistry .

Various techniques are available to decrease discomfort during LA injections. Transcutaneous electrical nerve stimulation (TENS) works on the principle of gate control theory. Transcutaneous electrical nerve stimulation directly stimulates the nerves by electrical impulses of short duration and small amplitude for pain reduction during LA injections . Transcutaneous electrical nerve stimulation proved to be more comfortable and beneficial in reducing pain and anxiety during LA injections.

Studies have reported that it lowers edema, nerve conduction velocities, cellular metabolism, and local blood flow .

Topical anesthetic agents are commonly used before the administration of LA . 2% lignocaine gel produces surface anesthesia; however, it has a limited capacity of penetrating deep into tissues. A cutaneous topical anesthetic which was first used in dermatology in the 1980s, Another recommended method to eliminate the pain of injection is cooling of the injection site. This technique has been used in sprains, burns, fractures, bruises, insect bites, and sports injuries

eutectic mixture of lignocaine and prilocaine (EMLA) - "a 1:1 mixture of 2.5% prilocaine and 2.5% lidocaine". The first trial to administer EMLA cream in the mucosal surface was first described by Holst and Evers.

ELIGIBILITY:
Inclusion Criteria:

* Class I and Class II relaying on ASA classification
* Children of the age-group 6-10 years were included in this study.
* Children who are never exposed to TENS, EMLA jelly,
* Children who require LA injections and in whom parental consent was obtained.
* Patients requiring LA for dental procedures such as pulpotomy, or extraction procedure.
* Definitely positive on frankel scale.

Exclusion Criteria:

* Children with epileptic disorder.
* Children with a history of cardiac and bleeding disorder.
* Immature children who cannot understand the concept of pain.
* Physically and mentally challenged children.
* Subjects allergic to LA drugs or cartridge components
* Patients having behavioral management problems.
* Patients having previous negative dental experience.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Baseline Heart Rate ( beats/min ) | mean measurement when the child is seated on the dental chair until right before the injection at 2 minute intervals. time frame was approximately Minute 0 - 2 ]
  Heart Rate will be measured by using digital manometerReading will be recorded at 2-minute intervals and the mean heart rate measurement will be calculated.
Heart Rate Measurement after Local Anaesthetic Administration( beats/min ) | After local anaesthetic solution delivery. Time frame is approximately minute 2 - 4
  Heart Rate will be measured by using digital manometer .Readings will be recorded at 2-minute intervals and the mean heart rate measurement will be calculated.
Baseline blood pressure systolic and diastolic ( mm Hg) | mean measurement when the child is seated on the dental chair until right before the injection at 2 minute intervals. time frame was approximately Minute 0 - 2 ]
  The blood pressure is most often measured in the arm when the patient is seated. Blood pressure readings taken in supine position tend to be lower than those taken in sitting position. Standards for blood pressure readings are based upon the seated position using the right arm.
Blood pressure measurment (systolic and diastolic)after local anesthetic administration ( mm Hg ) | After local anaesthetic solution delivery. Time frame is approximately minute 2 - 4
  The blood pressure is most often measured in the arm when the patient is seated. Blood pressure readings taken in supine position tend to be lower than those taken in sitting position. Standards for blood pressure readings are based upon the seated position using the right arm.
The FLACC scale or Face, Legs, Activity, Cry, Consolability scale | Approximately 2-4 minute after injection.
  The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Wong-Baker Faces Pain Rating Scale | Approximately 2-4 minute after injection.
  The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Bahy Ibarhim Abdelfatah, Principal Investigator — Minia University
Locations (1):
- El Minia university, Minya, Egypt